CLINICAL TRIAL: NCT04369534
Title: Efficacy and Safety of Individualized P2Y12 Receptor Antagonists Treatment Based on Agregometry Versus Fixed Dose Regimen in Patients After Acute Myocardial Infarction
Acronym: SPARELIFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: Croatian Science Foundation (Other Government); Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Davor Milicic, Professor Davor Milicic, MD, PhD, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8403
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Acute Coronary Syndrome; STEMI; NSTEMI - Non-ST Segment Elevation MI; PLATELET AGGREGATION; INDIVIDUALIZED THERAPY
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (Active Comparator): The patients randomized into the first group will be given the newer P2Y12 receptor inhibitor ticagrelor during the 12 months.
  Interventions: Drug: Ticagrelor
- Second group (Active Comparator): The second group of patients will be given ticagrelor initially, and after the first 30 days it will be replaced with clopidogrel, that will be given for the remaining time period (up to 12 months). Clopidogrel dosing will be modified according to the results of the aggregometry using the ADP test.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Adjusting clopidogrel dosage according to platelet reactivity results during 12 months after PCI
  Arms: Second group
Drug: Ticagrelor — Administration of standard dose of ticagrelor during 12 months after PCI
  Arms: First group

SUMMARY:
The specific goal of this study is to determine whether the individualized approach and adjusting the dosage of the P2Y12 receptor inhibitors will improve the platelet inhibiton and the clinical outcome in patients with an ACS, that were treated with PCI and the aforementioned drugs, but with an increased initial residual platelet activity. It is expected that the patients that have undergone the P2Y12 inhibitor therapy adjustment (according to the platelet reactivity measured by POC devices) will have better clinical outcomes (ie less ischemic events, without a significant increase in bleeding events) than those who did not undergo the therapy adjustment.

DETAILED DESCRIPTION:
In this study we plan to continue our previous research on individualized approach to platelet aniaggregation therapy in patients with an ACS treated with a PCI. The subjects included in this study will be adult patients successfully treated in our department for ACS (unstabile angina pectoris, non-ST segment elevation myocardial infarction and ST segment elevation myocardal infarction) with a PCI, a coronary stent implantation and the subsequent dual platelet antiaggregation therapy combining ASA and a P2Y12 receptor inhibitor. The diagnosis of different types of ACS will be made depending on the clinical presentation, ECG findings and changes in cardiac biomarker serum levels (troponin T and MB creatinine kinase isoezyme). Percutaneous coronary revascularization and the dual platelet antiaggregation therapy are the basis of the modern ACS treatment. Because the newer P2Y12 receptor inhibitors are not momentarily widely available in Croatia, the initial treatment will include the combination of ASA and clopidogrel. The exclusion critera are as following: postinterventional continuous GPIIb/IIIa inhibitor therapy, thrombocytopenia (<150x10E9/L), signifcant renal failure (creatinine>200 µmol/L), anemia (Htc<30%), hemorrhagic diathesis, history of recent hemorrhagic or ischemic CVI (within 6 months of admission), recent surgical procedure (within 6 weeks of admission) and an indication for chronic anticoagulant therapy. Also patients older than 80 years of age will not be included into this study. The necessary number of subjects is between 100 and 120.

Aggregometry using the ADP test will be done to all the patients without the exclusion criteria that were successfully treated wth PCI. The testing will be done within 24 hours of the intervention in order to determine the pharmacodynamic effect P2Y12 receptor inhibitors have on platelets and their reactivity. The optimal platelet reactivity (according to the international consensus) is between 19 and 46 U (49). The patients that will have an increased residual PR (>46 U) after being given the loading doses of clopidogrel will be included in this study and randomized into three groups using a computer software (Research Randomizer). The patients randomized into the first group will be given the newer P2Y12 receptor inhibitor ticagrelor during the 12 months. The second group of patients will be given ticagrelor initially, and after the first 30 days it will be replaced with clopidogrel, that will be given for the remaining time period (up to 12 months). Clopidogrel dosing will be modified according to the results of the aggregometry using the ADP test. The third group of patients will have the same therapy regiment as the second group, but will be given the standard doses of clopidogrel regardless of the aggregometry findings. The follow-up period, during which the dual platelet antiaggregation therapy will be administered, is going to be 12 months for each patient. Within this time-frame, total of ten PR measurements will be done. The measurements in the first month are scheduled as follows: on the first, second, third, seventh and thirtieth day after the ACS and the PCI. The following measurements are scheduled two, three, six, nine and twelve months after the ACS and the PCI.

ELIGIBILITY:
Inclusion Criteria:

* STEMI
* NSTEMI
* Unstable Angina
* Successful PCI
* Signed informed consent

Exclusion Criteria:

* >80 years of age at time of inclusion
* Cardiogenic shock
* Unsuccessful PCI
* GI bleed within the last 6 months
* Hemorrhagic CVI within last 6 months
* Ischemic CVI within last 6 months
* Major surgery within last 6 months
* Malignant disease
* Platelet count <=150
* Hematocrit <=30% or >=52%
* Creatinine >=200
* Chronic anticoagulant therapy
* Thrombotic thrombocytopenic purpura, leukemia, myelodysplasia
* Other: did not sign informed consent, refused, lives far away, leading physician doesn't want the patient to take part or any other reason leading to not signing the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ischemic events | During 1 year of follow up
  rehospitalization due to myocardial ishemia, another PCI, non-fatal acute myocardial infarction, "in-stent" thrombosis, transient ischemic attack (TIA), cerebrovascular insult (CVI) and cardiovascular death
Incidence of Hemorrhagic events | During 1 year of follow up
  Hemorrhagic events will be classified according to the BARC system, which represents an international consensus on documenting and classifying these events in cardiologic studies.
MACCE | During 1 year of follow up
  Data concerning mortality and other adverse cardiac and cerebrovascular events (MACCE) will be verified by examining the medical records. If no other cause of death was verified or documented, each fatal event will be regarded as being of cardiac etiology.

CONTACTS AND LOCATIONS:
Locations (1):
- Uhiversity hospital Center Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No